CLINICAL TRIAL: NCT00174668
Title: 52-week, Open, Randomized, Multinational, Multicenter Clinical Trial Comparing Insulin Glulisine in Combination With Insulin Glargine in an Intensified Insulin Regimen to a Two-injection Conventional Insulin Regimen in Type 2 Diabetes Mellitus Patients With Poor Glycemic Control Pretreated With a Two-injection Conventional Insulin Therapy
Brief Title: Insulin Glulisine in Diabetes Mellitus, Type 2
Acronym: GINGER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMR1964A_3504; EUDRACT # : 2004-001287-49
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin glulisine; Convulsive Therapy; Insulin Glargine

ARMS (2):
- 1 (Experimental): Mealtime insulin glulisine 3x daily and insulin glargine 1 x daily subcutaneously
  Interventions: Drug: Insulin Glulisine; Drug: Insulin Glargine
- 2 (Active Comparator): Two daily injection conventional insulin therapy
  Interventions: Drug: Insulin Therapy

INTERVENTIONS:
Drug: Insulin Glulisine — insulin glulisine 3 x daily (TID) subcutaneously 15 min before the start of a meal
  Arms: 1
Drug: Insulin Therapy — NPH (70%) plus regular insulin or insulin aspart (30%)
  Arms: 2
Drug: Insulin Glargine — 1 x daily (OD) subcutaneously at any time (but every day at the same time) according to BG
  Arms: 1

SUMMARY:
Primary objective:

The primary study objective is to demonstrate superior efficacy of an intensified insulin regimen with insulin glulisine and insulin glargine to a two-injection conventional insulin regimen in terms of change in glycated hemoglobin A1c (HbA1c), from baseline to endpoint.

Secondary objectives:

Secondary study objectives are to compare the intensified insulin regimen with insulin glulisine and insulin glargine to a two-injection conventional insulin regimen in terms of blood glucose (BG) values (fasting, pre-/postprandial (ppBG), nocturnal, mean daily, fasting plasma glucose), daily BG profiles, BG and HbA1c response rates (predefined), hypoglycemic events, adverse events, change of late diabetes complications, weight, body-mass-index, course of total daily insulin dose and adjustment, blood lipid profile, microalbuminuria, standard lab and quality of life/treatment satisfaction.

ELIGIBILITY:
Inclusion criteria :

Subjects meeting all of the following criteria will be considered for enrollment into the study:

* Type 2 diabetes mellitus, as defined by the American Diabetes Association for at least five years, treated with insulin for at least 6 months (no history of ketoacidosis).
* HbA1c between 7.5% and 11.0%, inclusive at both pre-screening and pre-randomization (week -2).
* For at least 3 months prior to week -8 visit, subjects must have been on a stable insulin regimen with two daily s.c. injections of premixed insulin: NPH plus regular insulin or NPH plus rapid acting insulin (insulin lispro or insulin aspart) in a mixture of 70/30 or 75/25. "Stable" means no change in regimen and no more than 30 % change in dose. Optionally, the subject can have been treated in addition with metformin according to its current official product information leaflet, treatment with other oral blood glucose lowering drugs is not allowed.
* Documentation of a full ophthalmologic exam (incl. fundoscopy)during the 6 months prior to randomization.
* Women are either not of childbearing potential (surgically sterile, or postmenopausal for more than 2 years). Women of childbearing potential must not be pregnant and agree to use a reliable contraceptive measure for the duration of the study. Reliable contraceptive measures include the following: systemic contraceptive (oral, implant, injections), diaphragm with intravaginal spermicide, cervical cap, intrauterine device or condom with spermicide.
* Willing and able to perform specified home blood glucose monitoring and to otherwise comply with study protocol requirements.
* Willing to change from a twice daily insulin regimen to a regimen requiring four daily insulin injections.
* Provision of signed and dated informed consent prior to any study procedures."Prescreening" informed consent, obtained in writing for all subjects, may be used during screening, but full study-specific informed consent must be obtained in writing for all subjects after any post-screening procedures.

Exclusion criteria :

Subjects presenting with any of the following will not be included in the study:

* Two or more severe hypoglycemic episodes within the past 3 months, or any hospitalization or emergency room visit due to poor diabetic control within the past 3 months prior to randomization.
* History of hypoglycemia unawareness.
* Impaired hepatic function, as shown by, but not limited to, ALAT (SGPT) or ASAT (SGOT) above 2x the upper limit of normal as measured at visit 1.
* Impaired renal function, as shown by, but not limited to, serum creatinine > 177 mmol/l (> 2 mg/dl) as measured at visit 1 (if no lower values due to individual metformin intake are required) or current renal dialysis.
* Body mass index (BMI) > 38 kg/m2.
* Any other clinically significant abnormalities on screening laboratory evaluation (unless discussed with the monitor and approved by the study management).
* Active proliferative diabetic retinopathy, as defined by the application of focal or panretinal photocoagulation or vitrectomy, in the 6 months prior to visit 1, or any other unstable (rapidly progressing) retinopathy that may require surgical treatment (including laser photocoagulation) during the study.
* History of hypersensitivity to insulin or insulin analogues or any of the excipients in the HMR 1964 formulation.
* Donation of blood or transfusion during the 2 months prior to the screening visit.
* Pregnant or lactating women, or women planning to become pregnant during the study.
* Treatment with any investigational drug in the last month before visit 1 (screening).
* Mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the study.
* Any clinically significant major organ system disease such as relevant cardiovascular, gastrointestinal, hepatic, neurologic, endocrine, hematologic or other major systemic diseases making implementation of the protocol or interpretation of the study results difficult.
* Treatment or likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol.
* History of drug or alcohol abuse within the last 2 years or current addiction to substances of abuse.
* Night shift workers.
* Subject unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study.
* Subject is the investigator or any subinvestigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2004-11; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
HbA1c | From baseline to study endpoint
Self monitored BG (SMBG) values | During the whole treatment phase
Body weight/body mass index (BMI) | From baseline to study endpoint and all other visits
Fasting blood lipid profile | From baseline to study endpoint and all other visits
Urine albumin | From baseline to study endpoint and all other visits
Total daily insulin dose | From baseline to study endpoint

SECONDARY OUTCOMES:
Adverse events | Throughout the study,
Standard laboratory tests | From baseline to study endpoint and all other visits
Vital signs | From baseline to study endpoint and all other visits
Physical examination | From baseline to study endpoint and all other visits

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Pilorget, MD, Study Director — Sanofi
Locations (15):
- Sanofi-Aventis, North Ryde, Australia
- Sanofi-Aventis, Brussels, Belgium
- Sanofi-Aventis, Prague, Czechia
- Sanofi-Aventis, Paris, France
- Sanofi-Aventis, Berlin, Germany
- Sanofi-Aventis, Milan, Italy
- Sanofi-Aventis, Gouda, Netherlands
- Sanofi-Aventis, Warsaw, Poland
- Sanofi-Aventis, Porto Salvo, Portugal
- Sanofi-aventis, Bucharest, Romania
- Sanofi-Aventis, Bratislava, Slovakia
- Sanofi-Aventis, Barcelona, Spain
- Sanofi-Aventis, Stockholm, Sweden
- Sanofi-Aventis, Meyrin, Switzerland
- Sanofi-Aventis, Guildford, United Kingdom

REFERENCES:
- [Derived] Fritsche A, Hahn A, Landgraf W, Haring HU. Incidence of Hypoglycaemia in Patients with Type 2 Diabetes - A Subgroup Analysis from the GINGER study. Eur Endocrinol. 2013 Mar;9(1):1-3. doi: 10.17925/EE.2013.09.01.1. Epub 2013 Apr 4. PMID 30349602